CLINICAL TRIAL: NCT03995979
Title: Short-Term Dietary Protein Restriction Modulation of Skeletal Muscle Bioenergetics and Innate Immunity
Brief Title: Inflammation and Protein Restriction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Malcom Randall VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB201900988 -V; NF/SGVHS (Other: Malcom Randall VA Medical Center)
Record Dates: First submitted 2019-06-21; First posted 2019-06-24 (Actual); Results first posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Protein Restriction; Diet; Inflammation
MeSH Terms: conditions — Inflammation | interventions — Diet, Protein-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Protein Restriction Group (Experimental): Subjects will follow a 4 day protein restricted diet using Scandishake® mixed with almond milk which will be provided.
  Interventions: Other: 4 Day Protein Restricted Diet

INTERVENTIONS:
Other: 4 Day Protein Restricted Diet — Subjects will follow a 4 day protein restricted diet using Scandishake® mixed with almond milk which will be provided. They may also drink water. No food, other beverages, or alcohol may be consumed. The amount of diet to be consumed will be calculated for each patient based upon resting energy expenditures plus additional energy needs. These will be consumed by the study subjects at home in an unrestricted manner, in that they may be consumed at any point of time in the day.
  Other Names: Scandishake

SUMMARY:
There is strong scientific data that supports that short-term protein restrictive diets reduce surgical stress responses. The investigators are hoping to use the information collected from the blood serum and muscle tissue of healthy subjects to help understand the baseline and early changes in muscle energetic and cell-mediated inflammation. The study team hopes to use the data collected in this pilot study to compare with patients undergoing open abdominal aortic aneurysm (AAA) repair in a future study

DETAILED DESCRIPTION:
Modulation of a patient's diet, specifically via short-term dietary protein restriction, can impact changes in cell energetics and dampen the normal subclinical inflammatory state. These changes can provide benchmarks for future research focused on using nutritional interventions aimed at improving the probability of a successful outcome following open aortic aneurysm surgery. The investigators will conduct a short term dietary restriction protocol to characterize these changes in a normal control cohort to be compared to patients which undergo surgery, to identify the optimal time points for sampling in the surgical population. These changes will be characterized by looking at inflammatory cells in the blood, proteins excreted in the urine, changes in microbiome signature identified by stool sample and oral swab, as well as changes in muscle energetics in small muscle biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers between 18 and 70 years of age

Exclusion Criteria:

* Age less than 18 years.
* The presence of any significant medical condition that might significantly confound the collection of biological data in the study including cancer, diabetes, inflammatory bowel disease (IBD), Advanced Renal Disease, Nut Allergy
* Unwilling to follow protocol
* Participation in another interventional clinical trial.
* Prisoners, pregnancy, or direct employees of the investigative team

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2024-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Scali, MD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - Malcom Randall VA Medical Center, Gainesville, Florida
  - UF Health---Vascular Surgery, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy, young adult males and females free of chronic medical conditions were recruited to participate in this study. Informed consent was obtained from all subjects before study participation, and this study was approved by the University of Florida's institutional review board (UF IRB#201900988). Advertisements were created for the general public for recruitment of participants with no clinical relationship.
Pre-assignment Details: Of 12 enrolled participants, 10 met inclusion criteria and commenced study intervention.
Period: Overall Study
Arm/Group | Protein Restriction Group
Started | 12
Completed | 10
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: 10 healthy individuals were recruited to participate in the study: five males and five females. Originally, 12 participants in total agreed to participate in the study following completion of the informed consent form, but two were withdrawn before the study procedural commenced.
Arm/Group | Protein Restriction Group
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants] — Population: 10 healthy individuals were recruited to participate in the study: five males and five females. Originally, 12 participants in total agreed to participate in the study following completion of the informed consent form, but two were withdrawn before the study procedural commenced.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 10
    >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.2 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 10 healthy individuals were recruited to participate in the study: five males and five females. Originally, 12 participants in total agreed to participate in the study following completion of the informed consent form, but two were withdrawn before the study procedural commenced.
  Participants
    Female | 5
    Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 10 healthy individuals were recruited to participate in the study: five males and five females. Originally, 12 participants in total agreed to participate in the study following completion of the informed consent form, but two were withdrawn before the study procedural commenced.
  Participants
    Hispanic or Latino | 1
    Not Hispanic or Latino | 9
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 10 healthy individuals were recruited to participate in the study: five males and five females. Originally, 12 participants in total agreed to participate in the study following completion of the informed consent form, but two were withdrawn before the study procedural commenced.
  Participants
    American Indian or Alaska Native | 0
    Asian | 2
    Native Hawaiian or Other Pacific Islander | 1
    Black or African American | 0
    White | 6
    More than one race | 0
    Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants] — Population: 10 healthy individuals were recruited to participate in the study: five males and five females. Originally, 12 participants in total agreed to participate in the study following completion of the informed consent form, but two were withdrawn before the study procedural commenced.
  participants
    United States | 10
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] — Population: 10 healthy individuals were recruited to participate in the study: five males and five females. Originally, 12 participants in total agreed to participate in the study following completion of the informed consent form, but two were withdrawn before the study procedural commenced.
  kg/m2 | 24.7 (4.0)

OUTCOME MEASURES:

1. Primary Outcome: Changes in the Human Intestinal Microbiome That Result From Short Term Dietary Adjustment.
Description: Genomic sequencing along with taxonomic and functional pathways analysis is used to identify any compositional and functional changes in the intestinal microbiome of patients on short-term dietary restrictions in relation its anti-inflammatory effects on pre-operative conditioning,
Time Frame: Day 2; Day 4; Day 7
Measure: Number; unit: Number of immunity related genes
Arm/Group | Protein Restriction Group
Number analyzed (Participants) | 10
Number of immunity related genes
  Differential expression of genes on Day 2 of DR compared to baseline | 232
  Differential expression of genes on day 4 DR compared to baseline | 172
  Differential expression of genes on day 7 DR compared to baseline | 145
  Total genes upregulated on day 2 of DR | 93
  Total genes upregulated on day 4 of DR | 24
  Total genes upregulated on day 7 of DR | 85
  Total genes downregulated on day 2 of DR | 139
  Total genes downregulated on day 4 of DR | 148
  Total genes downregulated on day 7 of DR | 60
Statistical Analysis 1: Comparison: Protein Restriction Group; A compositional analysis with species-level alpha diversity will be performed between the three conditions (Pre-Dietary Restriction, Dietary Restriction, and Post-Dietary Restriction,) with ANOVA testing. Furthermore, a differential abundance analysis will be performed to further identify and confirm prevalent organisms associated with the experimental dietary restriction; Test type: Superiority; p = 0.05, Paired t-test — The P-value was calculated using a paired t test

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Protein Restriction Group
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
The specific diet used in this study,although advantageous for its feasibility in achieving the targeted percent protein goal and caloric restriction, may deviate from the ideal short-term protein-calorie dietary restriction (stDR). Moreover, observations could be attributed to the diet itself and not necessarily from protein or caloric restrictions. Lastly, this study lacks a description of the peripheral immune cell response.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-07-09): https://cdn.clinicaltrials.gov/large-docs/79/NCT03995979/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-20): https://cdn.clinicaltrials.gov/large-docs/79/NCT03995979/SAP_001.pdf
  • Informed Consent Form (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/79/NCT03995979/ICF_002.pdf